CLINICAL TRIAL: NCT04493671
Title: A Phase 1, Partially Blind, Placebo Controlled, Randomized, Combined Single Ascending Dose With a Food Effect Cohort, Multiple Ascending Dose, and Relative Bioavailability Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of TBAJ-876 in Healthy Adult Subjects
Brief Title: Evaluate Safety, Tolerability, PK of TBAJ-876 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Global Alliance for TB Drug Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TBAJ-876-CL-001
Record Dates: First submitted 2020-07-22; First posted 2020-07-30 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Pulmonary Disease; Tuberculosis, Pulmonary; Tuberculosis; Multi Drug Resistant Tuberculosis; Drug Sensitive Tuberculosis; Drug-resistant Tuberculosis; Mycobacterium Tuberculosis Infection
Keywords: TBAJ-876; Diarylquinoline; DARQ
MeSH Terms: conditions — Lung Diseases; Tuberculosis, Pulmonary; Tuberculosis; Tuberculosis, Multidrug-Resistant | interventions — TBAJ-876; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (16):
- TBAJ-876 10mg SAD (Active Comparator): Cohort 1 single dose of 10 mg TBAJ-876 (n=6) under fasted conditions
  Interventions: Drug: TBAJ-876 suspension
- TBAJ-876 25mg SAD (Active Comparator): Cohort 2, Single dose of 25 mg TBAJ-876 (n=6) under fasted conditions
  Interventions: Drug: TBAJ-876 suspension
- TBAJ-876 50mg SAD (Active Comparator): Cohort 3 single dose of 50 mg TBAJ-876 (n=6) under fasted conditions
  Interventions: Drug: TBAJ-876 suspension
- TBAJ-876 100mg fasted SAD (Active Comparator): Cohort 4, single dose of 100 mg TBAJ-876 (n=9) under fasted conditions
  Interventions: Drug: TBAJ-876 suspension
- TBAJ-876 100mg fed SAD (Active Comparator): Cohort 4, dose of 100 mg TBAJ-876 (n=10) under fed conditions
  Interventions: Drug: TBAJ-876 suspension
- TBAJ-876 200mg SAD (Active Comparator): Cohort 5 single dose of 200 mg TBAJ-876 (n=6) under fasted conditions
  Interventions: Drug: TBAJ-876 suspension
- TBAJ-876 400mg SAD (Active Comparator): Cohort 6, single dose of 400 mg TBAJ-876) (n=6) under fasted conditions
  Interventions: Drug: TBAJ-876 suspension
- TBAJ-876 800mg SAD (Active Comparator): Cohort 7, Single dose of 800 mg TBAJ-876 (n=6) under fasted conditions
  Interventions: Drug: TBAJ-876 suspension
- TBAJ-876 Placebo SAD (Placebo Comparator): Single dose matching placebo for TBAJ-876 under fasted conditions (n=13)
  Interventions: Drug: Placebo suspension
- TBAJ-876 25mg MAD (Active Comparator): 25 mg TBAJ-876 (n=9) for 14 days under fed conditions
  Interventions: Drug: TBAJ-876 suspension
- TBAJ-876 75mg MAD (Active Comparator): 75 mg TBAJ-876) (n=9) for 14 days under fed conditions
  Interventions: Drug: TBAJ-876 suspension
- TBAJ-876 200mg MAD (Active Comparator): 200 mg TBAJ-876 (n=9) for 14 days under fed conditions
  Interventions: Drug: TBAJ-876 suspension
- TBAJ-876 Placebo MAD (Placebo Comparator): Matching placebo for TBAJ-876 for 14 days under fed conditions (n=12)
  Interventions: Drug: Placebo suspension
- TBAJ-876 1x100 mg rBA fasted (Active Comparator): Single dose TBAJ-876 of 100 mg (1 x 100 mg tablet) (n=10) under fasted conditions
  Interventions: Drug: TBAJ-876 100 mg tablet
- TBAJ-876 1x100 mg rBA fed (Active Comparator): Single dose TBAJ-876 of 100 mg (1 x 100 mg tablet) (n=10) under fed conditions
  Interventions: Drug: TBAJ-876 100 mg tablet
- TBAJ-876 4x25 mg rBA fasted (Active Comparator): Single dose TBAJ-876 of 100 mg (4 x 25 mg tablets) (n=10) under fasted conditions
  Interventions: Drug: TBAJ-876 25 mg tablet

INTERVENTIONS:
Drug: TBAJ-876 suspension — TBAJ-876 oral suspension, orally administered
  Arms: TBAJ-876 100mg fasted SAD; TBAJ-876 100mg fed SAD; TBAJ-876 10mg SAD; TBAJ-876 200mg MAD; TBAJ-876 200mg SAD; TBAJ-876 25mg MAD; TBAJ-876 25mg SAD; TBAJ-876 400mg SAD; TBAJ-876 50mg SAD; TBAJ-876 75mg MAD; TBAJ-876 800mg SAD
Drug: Placebo suspension — Placebo for TBAJ-876 oral Suspension; orally administered
  Arms: TBAJ-876 Placebo MAD; TBAJ-876 Placebo SAD
Drug: TBAJ-876 100 mg tablet — TBAJ-876 100 mg tablets, orally administered
  Arms: TBAJ-876 1x100 mg rBA fasted; TBAJ-876 1x100 mg rBA fed
Drug: TBAJ-876 25 mg tablet — TBAJ-876 25 mg tablets, orally administered
  Arms: TBAJ-876 4x25 mg rBA fasted

SUMMARY:
A Phase 1, Partially Blind, Placebo Controlled, Randomized, Combined Single Ascending Dose (SAD) with a Food Effect Cohort (Part 1), Multiple Ascending Dose (MAD) (Part 2), and Relative Bioavailability (rBA) (Part 3) Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of TBAJ-876 in Healthy Adult Subjects

DETAILED DESCRIPTION:
This study is a three-part, partially blinded, placebo controlled, combined single ascending dose with food-effect, multiple ascending dose study, and a single dose relative bioavailability study conducted at one study center in the United States.

Safety will be assessed throughout the study for all subjects. Safety assessments will include physical examinations, vital signs, serial ECGs, cardiac monitoring, adverse events (AEs), and clinical laboratory tests (including hematology, serum chemistry, coagulation, and urinalysis).

ELIGIBILITY:
Key Inclusion Criteria:

All volunteers must satisfy the following criteria to be considered for study participation:

1. Is a healthy adult male or female, 19 to 50 years of age (inclusive) at the time of screening.
2. Has a body mass index (BMI) ≥18.5 and ≤32.0 (kg/m2) and a body weight of no less than 50.0 kg.
3. Is medically healthy with no clinically significant screening results (e.g., laboratory profiles normal or up to Grade 1 per DMID Toxicity Tables), as deemed by the Investigator.
4. Has not used tobacco- or nicotine-containing products (including smoking cessation products), for a minimum of 6 months before dosing.
5. If assigned to receive study drug under fed conditions, is willing and able to consume the entire high-calorie, high-fat breakfast meal in the timeframe required.

Key Exclusion Criteria:

1. History or presence of clinically significant cardiovascular (heart murmur), pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, psychiatric disease or any other condition that, in the opinion of the Investigator, would jeopardize the safety of the subject or the validity of the study results.
2. Any presence of musculoskeletal toxicity (severe tenderness with marked impairment of activity, or frank necrosis).
3. Has a positive test for hepatitis B surface antigen, hepatitis C antibody, or HIV at screening.
4. Current or history of prolonged QT syndrome15. Family history of long-QT syndrome or sudden death without a preceding diagnosis of a condition that could be causative of sudden death (such as known coronary artery disease, congestive heart failure, or terminal cancer).
5. If assigned to the fasted/fed cohort, is lactose intolerant.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 137 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Related Adverse Events in Part 1, Single Ascending Dose | Day 1 to Day 28
  Subjects will be monitored for any adverse events from the signing of the consent form until the end-of-study visit. The Investigator or a Sub-Investigator will assess its relationship to the study drug.
Number of Participants with Treatment-Related Adverse Events in Part 2, Multiple Ascending Dose | Day 1 to Day 133
  Subjects will be monitored for any adverse events from the signing of the consent form until the end-of-study visit. The Investigator or a Sub-Investigator will assess its relationship to the study drug.
Number of Participants with Treatment-Related Adverse Events in Part 3, Relative Bioavailability Study | Day 1 to Day 21
  Subjects will be monitored for any adverse events from the signing of the consent form until the end-of-study visit. The Investigator or a Sub-Investigator will assess its relationship to the study drug.

SECONDARY OUTCOMES:
AUCExtrap [Pharmacokinetic Analysis] | Days 1 - 28
  PK parameters will be calculated from plasma concentrations of TBAJ-876 TBAJ-876, M2, and M3. AUCExtrap is the percentage of AUCinf based on extrapolation.
AUCinf [Pharmacokinetic Analysis] | Days 1 - 28
  PK parameters will be calculated from plasma concentrations of TBAJ-876 TBAJ-876, M2, and M3. AUCinf is area under the concentration-time curve from time-zero extrapolated to infinity.
AUClast [Pharmacokinetic Analysis] | Days 1 - 28
  PK parameters will be calculated from plasma concentrations of TBAJ-876 TBAJ-876, M2, and M3. AUClast area under the concentration-time curve from time-zero to the time of the last quantifiable concentration; calculated using the linear trapezoidal rule.
AUCtau [Pharmacokinetic Analysis] | Days 1 - 28
  PK parameters will be calculated from plasma concentrations of TBAJ-876 TBAJ-876, M2, and M3. AUCtau is area under the concentration-time curve during the dosing interval; calculated using the linear trapezoidal rule.
Cavg [Pharmacokinetic Analysis] | Days 1 - 28
  PK parameters will be calculated from plasma concentrations of TBAJ-876 TBAJ-876, M2, and M3. Cavg is average concentration during the dosing interval.
Clast [Pharmacokinetic Analysis] | Days 1 - 28
  PK parameters will be calculated from plasma concentrations of TBAJ-876 TBAJ-876, M2, and M3. Clast is the last quantifiable concentration determined directly from individual concentration-time data.
CL/F [Pharmacokinetic Analysis] | Days 1 - 28
  PK parameters will be calculated from plasma concentrations of TBAJ-876 TBAJ-876, M2, and M3. CL/F is apparent total clearance after single administration.
CLss/F [Pharmacokinetic Analysis] | Days 1 - 28
  PK parameters will be calculated from plasma concentrations of TBAJ-876 TBAJ-876, M2, and M3. CLss/F is apparent total clearance after multiple administration.
Cmax [Pharmacokinetic Analysis] | Days 1 - 28
  PK parameters will be calculated from plasma concentrations of TBAJ-876 TBAJ-876, M2, and M3. Cmax is maximum concentration, determined directly from individual concentration-time data.
RAUC [Pharmacokinetic Analysis] | Days 1 - 28
  PK parameters will be calculated from plasma concentrations of TBAJ-876 TBAJ-876, M2, and M3. RAUC is accumulation factor during multiple dosing, based on AUCtau.
RCmax [Pharmacokinetic Analysis] | Days 1 - 28
  PK parameters will be calculated from plasma concentrations of TBAJ-876 TBAJ-876, M2, and M3. RCmax is accumulation factor during multiple dosing, based on Cmax.
Tlast [Pharmacokinetic Analysis] | Days 1 - 28
  PK parameters will be calculated from plasma concentrations of TBAJ-876 TBAJ-876, M2, and M3. Tlast is time of the last quantifiable concentration.
Tmax [Pharmacokinetic Analysis] | Days 1 - 28
  PK parameters will be calculated from plasma concentrations of TBAJ-876 TBAJ-876, M2, and M3. Tmax is time of the maximum concentration.
T1/2 [Pharmacokinetic Analysis] | Days 1 - 28
  PK parameters will be calculated from plasma concentrations of TBAJ-876 TBAJ-876, M2, and M3. T1/2 is the observed terminal half-life.
Vz/F [Pharmacokinetic Analysis] | Days 1 - 28
  PK parameters will be calculated from plasma concentrations of TBAJ-876 TBAJ-876, M2, and M3. Vz/F is apparent volume of distribution in the terminal phase.
λz [Pharmacokinetic Analysis] | Days 1 - 28
  PK parameters will be calculated from plasma concentrations of TBAJ-876 TBAJ-876, M2, and M3. λz is the observed terminal rate constant; estimated by linear regression through at least 3 data points in the terminal phase of the log concentration-time profile.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Lombardi, MD, Study Chair — Global Alliance for TB Drug Development
Locations (1):
- Worldwide Clinical Trials, San Antonio, Texas, United States

REFERENCES:
- [Result] Lombardi A, Pappas F, Nedelman J, Hickman D, Jaw-Tsai S, Olugbosi M, Bruinenberg P, Beumont M, Sun E. Pharmacokinetics and safety of TBAJ-876, a novel antimycobacterial diarylquinoline, in healthy subjects. Antimicrob Agents Chemother. 2024 Oct 8;68(10):e0061324. doi: 10.1128/aac.00613-24. Epub 2024 Aug 28. PMID 39194204

DOCUMENTS (2):
  • Study Protocol (2021-12-03): https://cdn.clinicaltrials.gov/large-docs/71/NCT04493671/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-25): https://cdn.clinicaltrials.gov/large-docs/71/NCT04493671/SAP_001.pdf